CLINICAL TRIAL: NCT06465992
Title: Single-Shot Liposomal Bupivacaine vs. Liposomal Bupivacaine Combined With Dexamethasone Prior to Foot and Ankle Procedures: A Prospective Randomized Controlled Trial
Brief Title: Liposomal Bupivacaine With Dexamethasone for Foot Surgery
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DPED20242471
Record Dates: First submitted 2024-06-14; First posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Foot Surgery; Ankle Surgery; Post Operative Pain; Popliteal Nerve Block
MeSH Terms: conditions — Pain, Postoperative | interventions — Injections; Bupivacaine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Study Group 1: Foot/Ankle Surgery with Exparel Nerve Block (Active Comparator): Prior to participants surgical procedure, the anesthesiologist will administer a popliteal and saphenous nerve block consisting of 20 mL Liposomal bupivacaine (Exparel) + 10 mL of 0.75% bupivacaine
  Interventions: Drug: Exparel 266 MG Per 20 ML Injection; Drug: Bupivacaine Hcl 0.75% Inj
- Study Group 2: Foot/Ankle Surgery with Exparel + Dexamethasone Nerve Block (Active Comparator): Prior to participants surgical procedure, the anesthesiologist will administer a popliteal and saphenous nerve block consisting of 20 mL Liposomal bupivacaine (Exparel) + 1 mL of 10 mg preservative free Dexamethasone + 10 cc's of 0.75% bupivacaine
  Interventions: Drug: Exparel 266 MG Per 20 ML Injection; Drug: Bupivacaine Hcl 0.75% Inj; Drug: Dexamethasone

INTERVENTIONS:
Drug: Exparel 266 MG Per 20 ML Injection — 20 mL Liposomal bupivacaine (Exparel, 266 mg) will be administered in the popliteal and saphenous block
Drug: Bupivacaine Hcl 0.75% Inj — 10 mL of 0.75% bupivacaine will be administered in popliteal and saphenous block
Drug: Dexamethasone — 1 mL of 10 mg Dexamethasone will be administered in the popliteal and saphenous block
  Arms: Study Group 2: Foot/Ankle Surgery with Exparel + Dexamethasone Nerve Block

SUMMARY:
This study aims to understand the ideal formulation to utilize in saphenous nerve and popliteal nerve blocks for foot and ankle procedures. It will examine the use of liposomal bupivacaine alone or liposomal bupivacaine with dexamethasone prior to foot and ankle procedures in peripheral nerve blocks. We will compare liposomal bupivacaine (Exparel) and liposomal bupivacaine (Exparel) combined with dexamethasone to determine if the addition of dexamethasone significantly decreases postoperative narcotic use and prolongs analgesic effects when administered in a popliteal and saphenous block prior to foot and ankle orthopedic procedures.

ELIGIBILITY:
Inclusion Criteria:

* Participants with foot and ankle procedures at Jefferson Surgery Center, Navy Yard
* Participants with foot and ankle orthopedic procedures requiring a preoperative nerve block
* Age 18 and older
* English speaking
* Ability to complete surveys by phone or in person
* Ability to provide informed consent

Exclusion Criteria:

* Revision foot and ankle cases
* Allergies to study medications
* Non-English speakers
* Known alcohol or narcotic abuse history
* Existing contract with a pain specialist due to underlying preoperative pain syndrome
* Preoperative opioid use within the 3 months prior to surgery
* Participants who are pregnant, plan to become pregnant, or are breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2024-06-17 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Amount of pain medication used after surgery | 14 days
  Collected as tablets taken since all participants will be prescribed oxycodone
Pain level after surgery | 14 days
  Participants will be asked daily what their pain levels are using the Visual Analog (VAS) pain scale

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedic Institute, Philadelphia, Pennsylvania, United States